CLINICAL TRIAL: NCT05036603
Title: Comparison of the Acute Effects of Chest Physiotherapy Methods Applied in Different Positions in Preterm Newborns
Acronym: therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanko University (Other)
Responsible Party: Principal Investigator, Hatice Adiguzel, PT, Assistant Proffessor, Sanko University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FTR
Record Dates: First submitted 2021-08-18; First posted 2021-09-05 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2022-08

CONDITIONS: Preterm Birth; Premature; Bronchopulmonary Dysplasia; Respiratory Distress Syndrome; Mechanical Ventilation Complication; Mechanical Ventilation Pressure High; Oxygen Toxicity; Neonatal Respiratory Failure; Atelectasis Neonatal; Pneumonia Neonatal; Lobar Collapse; Chronic Liver Disease; Hyaline Membrane Disease
Keywords: Newborn; preterm; chest physiotherapy; neonatal intensive care unit; mechanical ventilation
MeSH Terms: conditions — Premature Birth; Bronchopulmonary Dysplasia; Respiratory Distress Syndrome; Pulmonary Atelectasis; Hyaline Membrane Disease

STUDY DESIGN:
Intervention Model Description: 2 groups; different chest physitherapy approach and 1 grup(control): routine medical care for newborns and neonatal intensive care unit's routin daily care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 1/routin medical care and neonatal intensive care unit's daily care (No Intervention): Group 1 (n=20) routine medical treatment for newborns on mechanical ventilator respiratory support and CPAP; Appropriate antibiotics given according to the needs of the baby, enteral-parenteral nutrition, oral or nebulizer drugs for softening the secretion, vitamin supplements and routine nursing care will be provided.
- 2/active chest physiotherapy in modified drainage positions (Experimental): Group 2 (n=20) newborns on mechanical ventilator respiratory support and CPAP; A single session of active chest physiotherapy (CP) will be applied using modified drainage positions (avoiding the trendelenburg position, excessive position change and avoiding hand contact in babies younger than 30 weeks or who are sensitive to position change). Active CP in various modified drainage positions; It will consist of percussion and vibration methods with proprioceptive replacement stimulations. After these methods, aspiration will be performed and a suitable position will be given to the lobe that is desired to be ventilated. In addition, these patients will be given routine medical treatment consisting of appropriate antibiotics, enteral-parenteral nutrition, oral or nebulizer drugs for softening the secretion, vitamin supplements and routine nursing care.
  Interventions: Other: chest physiotherapy
- 3/active chest physiotherapy in prone positions (Experimental): Group 3 (n=20) newborns on mechanical ventilator respiratory support and CPAP; a single session of active chest physiotherapy treatment to be applied only in the prone position; Starting with proprioceptive stimulation, percussion and vibration methods will be applied. After these methods, aspiration will be performed and a suitable position will be given to the lobe that is desired to be ventilated. In addition, these patients will be given routine medical treatment consisting of appropriate antibiotics, enteral-parenteral nutrition, oral or nebulizer drugs for softening the secretion, vitamin supplements and routine nursing care.
  Interventions: Other: chest physiotherapy

INTERVENTIONS:
Other: chest physiotherapy — diffferent chest physiotherapy methods
  Arms: 2/active chest physiotherapy in modified drainage positions; 3/active chest physiotherapy in prone positions

SUMMARY:
Infants in the neonatal intensive care unit (NICU) may be lost due to risks such as being sensitive, frequent exposure to birth complications and being prone to infection. The most common causes of mortality in newborn babies in the world; Complications due to preterm delivery (28%), infections (26%) and perinatal asphyxia (23%) were reported. Respiratory problems are observed in 4-6% of newborns. These problems are also important causes of mortality in the neonatal period. Newborn infants are more likely to have respiratory distress due to difficulties in airway calibration, few collateral airways, flexible chest wall, poor airway stability, and low functional residual capacity.Invasive mechanical ventilation (IMV) is frequently used in the treatment of newborns with respiratory failure. Various ventilation modes and strategies are used to optimize mechanical ventilation and prevent ventilator-induced lung injury. Among the important issues to be considered in newborns connected to mechanical ventilator (MV); Choosing an appropriately sized endotracheal tube to reduce airway resistance and minimize respiratory workload, correct positioning, regular nursing care, chest physiotherapy, sedation-analgesia, and infection prevention are also included.

DETAILED DESCRIPTION:
Infants in the neonatal intensive care unit (NICU) may be lost due to risks such as being sensitive, frequent exposure to birth complications and being prone to infection. The most common causes of mortality in newborn babies in the world; Complications due to preterm delivery (28%), infections (26%) and perinatal asphyxia (23%) were reported. Respiratory problems are observed in 4-6% of newborns. These problems are also important causes of mortality in the neonatal period. Newborn infants are more likely to have respiratory distress due to difficulties in airway calibration, few collateral airways, flexible chest wall, poor airway stability, and low functional residual capacity.Invasive mechanical ventilation (IMV) is frequently used in the treatment of newborns with respiratory failure. Various ventilation modes and strategies are used to optimize mechanical ventilation and prevent ventilator-induced lung injury. Among the important issues to be considered in newborns connected to mechanical ventilator (MV); Choosing an appropriately sized endotracheal tube to reduce airway resistance and minimize respiratory workload, correct positioning, regular nursing care, chest physiotherapy, sedation-analgesia, and infection prevention are also included.The preference for using non-invasive mechanical ventilation (NIMV) modes in NICUs is also increasing. Despite this, the use of IMV is still often required in preterm infants in the need for respiratory support and in the treatment of respiratory failure. Today, extremely preterm infants are extubated quickly. Because prolonged IMV can be a very important risk factor in the development of Bronchopulmonary Dysplasia (BPD). The reason for this is the physiological characteristics of newborns such as airway maintenance and cleanliness, smaller airway calibration, reduction in collaterals, flexible chest wall, poor airway stability, and low functional residual capacity. A small amount of secretion in preterm infants can produce a large increase in airway resistance. This reduces airflow and without expiratory flow, secretions cannot be expelled. With chest physiotherapy (CP), adequate expiratory flow can be achieved without causing airway closure.Chest physiotherapy techniques (CP) create mechanical effects in the lung, increasing ventilation, facilitating the removal of secretions and preventing bronchial obstruction. This ensures correct protection of the airways and facilitates extubation. Prolonged intubation and increased length of stay in NICUs can also lead to complications such as atelectasis, respiratory infections and chronic lung disease. Decreased oxygenation and excessive accumulation of secretions cause widespread increase in airway resistance, leading to prolonged ventilation or oxygen support. Oxygen therapy is an integral part that is frequently used as respiratory support in NICUs. However, long-term oxygen therapy may cause excessive accumulation of bronchial secretions. This makes CP mandatory. Traditional CP has become an indispensable part of airway management in NICU settings to remove excess bronchial secretions and thereby increase oxygenation. There are many studies on CP in the literature.In some of these studies, it was found that it did not prevent atelectasis, that CP had no effect, or that CP accelerated weaning from MV. The role of CP in reducing respiratory morbidity in infants and neonates continues to be debated and more studies are needed. CP needs to be supported by well-controlled studies with large sample sizes, particularly regarding the techniques used and specific protocols. Therefore, in this study, it is aimed to compare the acute effects of CP methods applied in different positions in preterm newborns.

ELIGIBILITY:
Inclusion Criteria:

* Preterm newborns born <37 and >28 weeks due to MV or CPAP, hospitalized in the NICU and with a voluntary consent form from their families (with segmental lobar collapse as a result of Chest X-Ray, RDS/BPD/HMH/Atelectasis/Pneumonia/ Preterm newborns diagnosed with Chronic Pulmonary Disease or in stable condition with a thick and secretory focus on X-ray)
* First-time infants who have not received any chest physiotherapy program

Exclusion Criteria:

* Newborn infants who have been unstable in the last 2 days (SpO₂ <60 mmHg, heart rate, blood pressure, persistent apnea, excessive increases in respiratory rate, tachycardia, nasal wing breathing, cyanosis..etc)

  * Newborn infants with rib fracture, hemoptysis, diaphragmatic hernia, pulmonary hemorrhage, pneumothorax
  * Those diagnosed with any known heart disease or genetic disease
  * Those with osteopenia-osteoporosis or thrombocytopenia
  * Infants with any known neurological diagnosis (Abnormal MRI finding, Hydrocephalus, Chiari Malformation, Asphyxia, Periventricular Leukomolacia (PVL), Intraventricular Hemorrhage (IVH), Kernicterius, Hypoxic Ischemic Encephalopathy (HIE), Hydrocephalus)
  * Preterm infants weighing <1000 g
  * Infants born with congenital anomaly (Spina Bifida, Arthrogryposis Multiplex Congenita..etc)
  * Newborns undergoing any surgery

Ages: 1 Day to 45 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
heart rate | Before starting chest physiotherapy and up to15 minutes after ending therapy
  heart rate of the preterm newborns
chest X-Ray | on the 1st day before starting chest physiotherapy session and up to 24 hours after chest physiotherapy session
  chest X-Ray of the preterm newborns
arterial blood gases | on the 1st day before starting chest physiotherapy session and up to 24 hours after chest physiotherapy session
  arterial blood gases from the radial artery or from the umbilical catheter in infants with an umbilical catheter
PaO₂ | on the time before starting chest physiotherapy and up to 15 minutes after ending therapy
  PaO₂ of the preterm newborns
blood pressure | on the time before starting chest physiotherapy and up to15 minutes after ending therapy
  blood pressure of the preterm newborns
respiratory rate | Before starting chest physiotherapy and up to15 minutes after ending therapy
  respiratory rate of the preterm newborns
Peep (cm H₂O) | on the time before starting chest physiotherapy and up to 15 minutes after ending therapy
  Peep (cm H₂O) of the preterm newborns
Pip (cm H₂O) | on the time before starting chest physiotherapy and up to15 minutes after ending therapy
  Pip (cm H₂O) of the preterm newborns
FİO₂ (%/mm Hg) | on the time before starting chest physiotherapy and up to 15 minutes after ending therapy
  FİO₂ (%/mm Hg) of the preterm newborns
O₂ Saturation (mmHg) (SpO₂) | on the time before starting chest physiotherapy and up to 15 minutes after ending therapy
  O₂ Saturation (mmHg) (SpO₂) of the preterm newborns

SECONDARY OUTCOMES:
Chest shape and type (barrel/pektusexcavatum..etc) | on the time before starting chest physiotherapy and up to 15 minutes after ending therapy
  Chest shape and type (barrel/pektusexcavatum..etc) will be noted by inspection before and after chest physiotherapy.
Respiratory stress | before physiotherapy
  The chest will be inspected before physiotherapy to note any signs of respiratory stress (chest retraction, expiratory sound, wheezing, etc.) and skin color (cyanosis/pink-bright-vivid/pale-white).
the respiratory pattern | on the time before starting chest physiotherapy and up to 15 minutes after ending therapy
  Before and after chest physiotherapy, the physiotherapist will evaluate the respiratory pattern (tachypnea, periodic breathing, apnea, coughing, sneezing) by inspection.
Daily nutrition type | on the time before starting chest physiotherapy and up to 24 hours after chest physiotherapy
  Daily nutrition type will be learned and respiratory problems encountered during feeding will be learned from the nurse/mother and noted.

CONTACTS AND LOCATIONS:
Overall Officials: hatice Adiguzel, PhD, Principal Investigator — Kahramanmaras Sutcu Imam University
Locations (1):
- Kahramanmaras Sutcu Imam University, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
there is no plan to make individual participant data (IPD) available to other researchers.